CLINICAL TRIAL: NCT01930292
Title: A Phase I Study to Evaluate the Safety and Determine the Maximum Tolerated Dose (MTD) of Debio 1143 Combined With Carboplatin and Paclitaxel in Patients With Squamous Non-Small Cell Lung Cancer (NSCLC), Platinum-refractory Ovarian Cancer, and Basal-like/Claudin Low Triple Negative Breast Cancer (TNBC)
Brief Title: Debio 1143 in Combination With Carboplatin and Paclitaxel in Patient With Advanced Solid Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Part B was cancelled based on business decision
Sponsor: Debiopharm International SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Debio 1143-103; 2012-003676-40 (EudraCT Number)
Record Dates: First submitted 2013-06-21; First posted 2013-08-28 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-03

CONDITIONS: Solid Tumors
MeSH Terms: interventions — Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Part A: Debio 1143 (Experimental): Eligible participants receive Part A: Debio 1143 once daily for 5 consecutive days in each 21-day treatment cycle according to dose escalation rules (in combination with Paclitaxel and Carboplatin standard of care)
  Interventions: Drug: Part A: Debio 1143; Drug: Paclitaxel; Drug: Carboplatin
- Part B: Lung Cancer (Experimental): Participants with Lung Cancer receive Part B: Debio 1143 once daily for 5 consecutive days in each 21-day treatment cycle (in combination with Paclitaxel and Carboplatin standard of care)
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Part B: Debio 1143
- Part B: Ovarian Cancer (Experimental): Participants with Ovarian Cancer receive Part B: Debio 1143 once daily for 5 consecutive days in each 21-day treatment cycle (in combination with Paclitaxel and Carboplatin standard of care)
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Part B: Debio 1143
- Part B: Breast Cancer (Experimental): Participants with Breast Cancer receive Part B: Debio 1143 once daily for 5 consecutive days in each 21-day treatment cycle (in combination with Paclitaxel and Carboplatin standard of care)
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Part B: Debio 1143

INTERVENTIONS:
Drug: Part A: Debio 1143 — Adaptive doses of Debio1143 oral capsules, between 50 and 400 mg until the recommended dose (RD) is determined.
  Arms: Part A: Debio 1143
Drug: Paclitaxel — Paclitaxel standard of care, intravenous (IV), once on day 1 or 2 of each 21-day treatment cycle, after pre-medication to prevent severe hypersensitivity reactions.
Drug: Carboplatin — Carboplatin standard of care, intravenous (IV), once on day 1 or 2 of each 21-day treatment cycle.
Drug: Part B: Debio 1143 — RD of Debio1143 oral capsules, once daily for five consecutive days starting on day 1 or 2 of each 21-day treatment cycle.
  Arms: Part B: Breast Cancer; Part B: Lung Cancer; Part B: Ovarian Cancer

SUMMARY:
This is a two-part trial in patients with squamous non-small cell lung cancer (NSCLC), platinum (Pt)-refractory ovarian cancer, and basal-like/claudin low triple negative breast cancer (TNBC).

The primary objective of Part A is to determine the maximum tolerated dose (MTD) of Debio 1143 when administered to these patients in combination with full doses of paclitaxel and carboplatin.

The primary objective of Part B is to consolidate the safety profile of the recommended dose of Debio 1143 when administered to these patients in combination with full doses of paclitaxel and carboplatin.

ELIGIBILITY:
Inclusion Criteria:

* Meets protocol-specified criteria for qualification and contraception
* Is willing and able to remain confined in the study unit for the entire duration of each treatment period and comply with restrictions related to food, drink and medications
* Voluntarily consents to participate and provides written informed consent prior to any protocol-specific procedures

Exclusion Criteria:

* Has history or current use of over-the-counter medications, dietary supplements, or drugs (including nicotine and alcohol) outside protocol-specified parameters
* Has signs, symptoms or history of any condition that, per protocol or in the opinion of the investigator, might compromise:

  1. the safety or well-being of the participant or study staff;
  2. the safety or well-being of the participant's offspring (such as through pregnancy or breast-feeding); or
  3. the analysis of results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-04; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Part A: Number of participants with dose-limiting toxicities | up to 18 weeks
  Categories: each Debio 1143 dose level and overall
Part B: Percentage of participants with adverse events (AEs) and serious AEs (SAEs) according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) criteria | up to 18 weeks + 28 days

SECONDARY OUTCOMES:
Part A: Percentage of participants with AEs and serious adverse events (SAEs) according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) criteria | up to 18 weeks + 28 days
  Categories: each Debio 1143 dose level and overall
Part A: Number of participants with change in vital signs | up to 18 weeks
  Categories: each Debio 1143 dose level and overall
Part A: Number of participants with change in electrocardiogram (ECG) | up to 18 weeks
  Categories: each Debio 1143 dose level and overall
Part A: Number of participants with change in Eastern Cooperative Oncology Group (ECOG) performance status (PS) | up to 18 weeks
  Categories: each Debio 1143 dose level and overall
Part B: Number of participants with change in vital signs | up to 18 weeks
  Categories: each indication at the recommended dose (RD)
Part B: Number of participants with change in electrocardiogram (ECG) | up to 18 weeks
  Categories: each indication at the recommended dose (RD)
Part B: Number of participants with change in Eastern Cooperative Oncology Group (ECOG) performance status (PS) | up to 18 weeks
  Categories: each indication at the recommended dose (RD)
Part A: Percentage of participants with incidence of laboratory abnormalities according to NCI-CTCAE criteria | up to 18 weeks
  Categories: each Debio 1143 dose level and overall
Part B: Percentage of participants with incidence of laboratory abnormalities according to NCI-CTCAE criteria | up to 18 weeks
  Categories: each indication at the RD
Part A: Percentage of participants with treatment discontinuations due to AEs and SAEs | up to 18 weeks + 28 days
  Categories: each Debio 1143 dose level and overall
Part B: Percentage of participants with treatment discontinuations due to AEs and SAEs | up to 18 weeks + 28 days
  Categories: each indication at the RD
Part A: Number of participants with change in left ventricular ejection fraction (LVEF) | up to 18 weeks
  Categories: each Debio 1143 dose level and overall
Part B: Number of participants with change in left ventricular ejection fraction (LVEF) | up to 18 weeks
  Categories: each indication at the RD
Part A: Number of participants with tumour response: disease control, change in tumour size from baseline and overall response | up to 18 weeks
  Categories: each Debio 1143 dose level and overall
Part B: Number of participants with tumour response: disease control, change in tumour size from baseline and overall response | up to 18 weeks
  Categories: each indication at the RD
Part A: Percentage of participants with progression-free survival (PFS) at 6 months | at 6 months
  Categories: each Debio 1143 dose level and overall
Part B: Percentage of participants with progression-free survival (PFS) at 6 months | at 6 months
  Categories: each indication at the RD
Part A: Percentage of participants with survival at 1 year | at 12 months
  Categories: each Debio 1143 dose level and overall
Part B: Percentage of participants with survival at 1 year | at 12 months
  Categories: each indication at the RD
Part B: Maximum concentration (Cmax) in the pharmacokinetic (PK) subset | up to 18 weeks
  Categories: Debio 1143 alone; Debio 1143 when administered with paclitaxel and carboplatin; paclitaxel, 6αOH-paclitaxel (metabolite), and carboplatin (total and free Pt) when administered as chemotherapy alone; paclitaxel, 6αOH-paclitaxel (metabolite), and carboplatin (total and free Pt) when administered in combination with Debio 1143
Part B: Lowest concentration before the next dose (Ctrough) of Debio 1143 in the PK subset | up to 18 weeks
  Categories: alone and in combination with chemotherapy
Part B: Time to maximum concentration (tmax) in the PK subset | up to 18 weeks
  Categories: Debio 1143 alone; Debio 1143 when administered with paclitaxel and carboplatin; paclitaxel, 6αOH-paclitaxel (metabolite), and carboplatin (total and free Pt) when administered as chemotherapy alone; paclitaxel, 6αOH-paclitaxel (metabolite), and carboplatin (total and free Pt) when administered in combination with Debio 1143
Part B: Area under the concentration versus time curve from the beginning to a point in time (AUC0-t) in the PK subset | up to 18 weeks
  Categories: Debio 1143 alone; Debio 1143 when administered with paclitaxel and carboplatin; paclitaxel, 6αOH-paclitaxel (metabolite), and carboplatin (total and free Pt) when administered as chemotherapy alone; paclitaxel, 6αOH-paclitaxel (metabolite), and carboplatin (total and free Pt) when administered in combination with Debio 1143
Part B: Area under the concentration versus time curve extrapolated to infinity (AUC∞) in the PK subset | up to 18 weeks
  Categories: Debio 1143 alone; Debio 1143 when administered with paclitaxel and carboplatin; paclitaxel, 6αOH-paclitaxel (metabolite), and carboplatin (total and free Pt) when administered as chemotherapy alone; paclitaxel, 6αOH-paclitaxel (metabolite), and carboplatin (total and free Pt) when administered in combination with Debio 1143
Part B: Terminal rate constant (λz) in the PK subset | up to 18 weeks
  Categories: Debio 1143 alone; Debio 1143 when administered with paclitaxel and carboplatin; paclitaxel, 6αOH-paclitaxel (metabolite), and carboplatin (total and free Pt) when administered as chemotherapy alone; paclitaxel, 6αOH-paclitaxel (metabolite), and carboplatin (total and free Pt) when administered in combination with Debio 1143
Part B: Apparent terminal half-life (t½) in the PK subset | up to 18 weeks
  Categories: Debio 1143 alone; Debio 1143 when administered with paclitaxel and carboplatin; paclitaxel, 6αOH-paclitaxel (metabolite), and carboplatin (total and free Pt) when administered as chemotherapy alone; paclitaxel, 6αOH-paclitaxel (metabolite), and carboplatin (total and free Pt) when administered in combination with Debio 1143
Part B: Mean residence time (MRT) in the PK subset | up to 18 weeks
  Categories: Debio 1143 alone; Debio 1143 when administered with paclitaxel and carboplatin; paclitaxel, 6αOH-paclitaxel (metabolite), and carboplatin (total and free Pt) when administered as chemotherapy alone; paclitaxel, 6αOH-paclitaxel (metabolite), and carboplatin (total and free Pt) when administered in combination with Debio 1143
Part B: Apparent clearance (CL/F) of Debio 1143 in the PK subset | up to 18 weeks
  Categories: alone and in combination with chemotherapy
Part B: Apparent volume of distribution during the terminal phase (Vz/F) of Debio 1143 in the PK subset | up to 18 weeks
  Categories: alone and in combination with chemotherapy
Part B: Total amount of Debio 1143 excreted in urine (Ae) in the PK subset | up to 18 weeks
  Categories: alone and in combination with chemotherapy
Part B: Total amount of Debio 1143 excreted in urine in the first 8 hours (Ae0-8) in the PK subset | up to 18 weeks
  Categories: alone and in combination with chemotherapy
Part B: Total amount of Debio 1143 excreted in urine between 8 and 24 hours (Ae8-24) in the PK subset | up to 18 weeks
  Categories: alone and in combination with chemotherapy
Part B: Renal clearance calculated as Ae/AUC∞ (CLR) of Debio 1143 in the PK subset | up to 18 weeks
  Categories: alone and in combination with chemotherapy
Part B: Fraction of the dose excreted in urine calculated as Ae/dose (fe) of Debio 1143 in the PK subset | up to 18 weeks
  Categories: alone and in combination with chemotherapy
Part B: Area under the concentration versus time curve in the first 12 hours (AUC0-12) in the PK subset | up to 18 weeks
  Categories: paclitaxel, 6αOH-paclitaxel (metabolite), and carboplatin (total and free Pt) when administered as chemotherapy alone; paclitaxel, 6αOH-paclitaxel (metabolite), and carboplatin (total and free Pt) when administered in combination with Debio 1143
Part B: Total body clearance (CL) in the PK subset | up to 18 weeks
  Categories: paclitaxel, 6αOH-paclitaxel (metabolite), and carboplatin (total and free Pt) when administered as chemotherapy alone; paclitaxel, 6αOH-paclitaxel (metabolite), and carboplatin (total and free Pt) when administered in combination with Debio 1143
Part B: Volume of distribution at steady-state (Vss) in the PK subset | up to 18 weeks
  Categories: paclitaxel, 6αOH-paclitaxel (metabolite), and carboplatin (total and free Pt) when administered as chemotherapy alone; paclitaxel, 6αOH-paclitaxel (metabolite), and carboplatin (total and free Pt) when administered in combination with Debio 1143
Part B: Mean Residence Area under the concentration versus time curve (MR,AUC) in the PK subset | up to 18 weeks
  Categories: paclitaxel, 6αOH-paclitaxel (metabolite), and carboplatin (total and free Pt) when administered as chemotherapy alone; paclitaxel, 6αOH-paclitaxel (metabolite), and carboplatin (total and free Pt) when administered in combination with Debio 1143
Part B: Mean Residence Maximum Concentration (MR,Cmax) in the PK subset | up to 18 weeks
  Categories: paclitaxel, 6αOH-paclitaxel (metabolite), and carboplatin (total and free Pt) when administered as chemotherapy alone; paclitaxel, 6αOH-paclitaxel (metabolite), and carboplatin (total and free Pt) when administered in combination with Debio 1143
Part B: Platinum Refraction (PtR) in ovarian cancer participants included in the PK subset | up to 18 weeks
  Categories: paclitaxel, 6αOH-paclitaxel (metabolite), and carboplatin (total and free Pt) when administered as chemotherapy alone; paclitaxel, 6αOH-paclitaxel (metabolite), and carboplatin (total and free Pt) when administered in combination with Debio 1143
Part B: Cmax in patients other than the PK subset | up to 18 weeks
  Categories: paclitaxel, 6αOH-paclitaxel (metabolite), and carboplatin (total and free Pt) when administered as chemotherapy alone; paclitaxel, 6αOH-paclitaxel (metabolite), and carboplatin (total and free Pt) when administered in combination with Debio 1143
Part B: Concentration observed at time n (Cn) following Debio 1143 administration in patients other than the PK subset | up to 18 weeks
  Categories: paclitaxel, 6αOH-paclitaxel (metabolite), and carboplatin (total and free Pt) when administered as chemotherapy alone; paclitaxel, 6αOH-paclitaxel (metabolite), and carboplatin (total and free Pt) when administered in combination with Debio 1143

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre Delord, MD, Study Chair — Institut Claudius Regaud, Toulouse, France
Locations (4):
- France (4):
  - Centre Georges François Leclerc, Dijon
  - Centre Léon Bérard, Lyon
  - Institut Curie, Paris
  - Institut Claudius Regaud, Toulouse

REFERENCES:
- See also: Site Debiopharm SA — http://www.debiopharm.com